CLINICAL TRIAL: NCT02155803
Title: ACTHAR GEL for Sarcoidosis-Associated Calcium Dysregulation: An Open-label Pilot Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Marc A. Judson, MD, Marc A. Judson, MD, Albany Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCMAJCA2014
Record Dates: First submitted 2014-05-30; First posted 2014-06-04 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Sarcoidosis; Hypercalcemia Due to Sarcoidosis
Keywords: Sarcoidosis-Associated Calcium Dysregulation; Sarcoidosis-Associated hypercalciuria; hypercalcemia; hypercalciuria; nephrocalcinosis; nephrolithiasis; interstitial nephritis; glomerulonephritis; acute kidney disease; chronic kidney disease
MeSH Terms: conditions — Sarcoidosis; Hypercalcemia; Hypercalciuria; Nephrocalcinosis; Nephrolithiasis; Nephritis, Interstitial; Glomerulonephritis; Renal Insufficiency, Chronic | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sarcoidosis related Calcium Dysregulation (Experimental): Subjects with Sarcoidosis associated calcium dysregulation will be administered 80 units of Acthar Gel (adrenocorticotropic hormone) twice a week for 12 weeks. Clinical visits will be scheduled for -30 days, day of 1st dose and 4,8,12 and 16 week after 1st dose to monitor the health of subjects.
  Interventions: Drug: ACTHAR Gel (adrenocorticotropic hormone)

INTERVENTIONS:
Drug: ACTHAR Gel (adrenocorticotropic hormone) — ACTHAR GEL (adrenocorticotropic hormone) 80 units subcutaneously twice weekly for 12 weeks

SUMMARY:
ACTHAR Gel has activity in sarcoidosis associated hypercalciuria and calcium dysregulation.

DETAILED DESCRIPTION:
Sarcoidosis is a multisystem granulomatous disease of unknown cause. Although sarcoidosis most commonly affects the lung, it may affect any organ. Although corticosteroids are recognized as the drug of choice for sarcoidosis. ACTH(adrenocorticotropic hormone) is the only drug that is FDA-approved for this disorder. However, there is limited data on the efficacy of ACTH for this condition.

Calcium metabolism is disregulated in active sarcoidosis. The primary abnormality in calcium metabolism stems from an increased 1-α hydroxylase activity in sarcoid alveolar macrophages that converts 25-hydroxyvitamin D to 1, 25-dihydroxyvitamin D, the active form of the vitamin. This can result in hypercalcemia, hypercalciuria, nephrocalcinosis, nephrolithiasis, interstitial nephritis, glomerulonephritis, acute and chronic kidney disease. Importantly, almost of the renal manifestations stem from disordered calcium metabolism. Unlike other organ manifestations of sarcoidosis, the disorder of calcium metabolism is more common in whites compared to african americans.Compared to hypercalcemia, hypercalciuria is three times more common in sarcoidosis, nevertheless, it has largely been ignored.

In general, the patient with hypercalcemia should be advised to avoid sunlight, curtail intake of major sources of dietary calcium and vitamin D, and drink ample fluids.If the patient is symptomatic, serum calcium is greater than 11 mg/dl, the serum creatinine is elevated, or the patient has nephrolithiasis, drug therapy is usually required. The drug of choice is prednisone at an initial daily dose of 20 - 40 mg/day.Unfortunately, prolonged corticosteroid therapy may result in unacceptable side effects including osteoporosis. This is particularly important as elevated calcitriol observed in patients with sarcoidosis can further jeopardize bone structure by resorption. Alternative medications that have shown benefit for sarcoidosis associated calcium dysregulation have included chloroquine,hydroxychloroquine, ketoconazole.

Not only may ACTHER GEL have obvious anti-inflammatory effects by resulting in corticosteroid production, but it may also activate melanocortin receptors. The melanocortin system has powerful anti-inflammatory properties that may be beneficial in the treatment of sarcoidosis.

We believe that there are several specific advantages of assessing the effectiveness of anti-sarcoidosis therapy by examining sarcoidosis-associated disorders of calcium metabolism.

1. The measures of granulomatous activity (serum calcium, urinary calcium, serum 25-hydroxyvitamin D, and serum 1, 25-dihydroxyvitamin D levels) are directly related to the granulomatous inflammation of sarcoidosis.
2. These parameters can be accurately and objectively quantified. This is an important issue in sarcoidosis as the endpoint for involvement of the lungs, skin, and eyes is problematic because it is either inexact and/or not unidimensional.
3. These constituents can be easily used to clinically monitor sarcoidosis. This is not the case for other forms of sarcoidosis including involvement of the lung and skin.

   * Although hypercalciuria and disordered calcium metabolism is not as common a manifestation of sarcoidosis as lung involvement, there is little evidence that the anti-granulomatous response to this disease is organ specific. In a randomized double-blind placebo control trial of infliximab for pulmonary sarcoidosis, extrapulmonary sarcoidosis also responded to this therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years old.
2. Able to understand English to the point of comprehending the informed consent form.
3. Biopsy proven sarcoidosis.
4. Documented hypercalciuria (urinary excretion of > 4mg/kg of calcium/day) or hypercalcemia within 4 weeks of study entry.
5. Historical evidence that the patient's hypercalciuria/hypercalcemia is related to sarcoidosis. This should include a serum parathyroid hormone (PTH) level which is not elevated.

Exclusion Criteria:

1. A change in anti-sarcoidosis medications within 3 months of study entry.
2. A history of hyperparathyroidism or another non-sarcoidosis cause of hypercalcemia/hypercalciuria
3. A history of Cushing's disease.
4. Have a diagnosis of a medical disorder other than sarcoidosis that in the opinion of the investigator would complicate the evaluation of response treatment.
5. Have used any investigational drug within 1 month prior to screening or within 5 half-lives of the investigational agent, whichever is longer.
6. Use of loop or thiazide diuretics for hypertension or other disorders.
7. Chronic use of antacids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Reduction of 24 hour urine calcium | Between week 0 and week 12.
  Reduction of 24 hour urine calcium in patients with sarcoidosis associated hypercalciuria (primary endpoint) between week 0 and week 12.

SECONDARY OUTCOMES:
Change in serum calcium during 12 week ACTHAR GEL treatment | Baseline compared to 12 weeks.
Change in 1,25 di-hydroxy Vitamin D during 12 week ACTHAR GEL treatment | Baseline compared to 12 weeks.
Change in patient global VAS during 12 week ACTHAR GEL treatment | Baseline to 12 weeks
Change in physician global VAS during 12 week ACTHAR GEL treatment | Baseline to 12 Weeks
Change in urinary symptoms during 12 week ACTHAR GEL treatment | Baseline to 12 Weeks
Change in Short Form-36 during 12 week ACTHAR GEL treatment | Baseline to 12 Weeks
Change in Sarcoidosis Health Questionnaire during 12 week ACTHAR GEL treatment | Baseline to 12 Weeks
Change in eCOST during 12 week ACTHAR gel treatment | Baseline to 12 Weeks
Change in adjusted eCOST (eCOSTadj) calculated as the eCOST/# organs with an eCOST score > 022 during 12 week ACTHAR gel treatment | Baseline to 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Judson, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical College, Albany, New York, United States